CLINICAL TRIAL: NCT00369213
Title: Randomised Controlled Trial of the Effect of Additional Spermicidal Lubrication on Condom Failure
Brief Title: Randomised Controlled Trial of Condoms Plus Additional Lubrication
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Manchester (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: RDO/18/67
Record Dates: First submitted 2006-08-24; First posted 2006-08-29 (Estimated); Last update posted 2006-08-29 (Estimated); Status verified 2004-12

CONDITIONS: Contraception
Keywords: Crossover trial; condom failure; additional spermicidal lubricant

INTERVENTIONS:
Device: Additional spermicidal lubricant to condoms

SUMMARY:
This RCT compares the clinical and non clinical condom failure rate among condom using heterosexual couples with and without externally applied additional spermicidal lubricant. The hypothesis is that breakage and slippage rates will be reduced.

DETAILED DESCRIPTION:
A recent retrospective cohort study of 1006 subjects reported a marked reduction in condom failure amongst users applying additional lubrication. Improving the reliability of condoms would reduce the incidence of unwanted pregnancies and STI's (and hence health and social costs). This trial investigates the relative risk reduction amongst couples applying additional spermicidal lubrication to condoms, other factors associated with condom failure, the acceptability and side effects of additional spermicide and its cost effectiveness.

200 regular condom users will be recruited from family planning clinics and other community sources. A randomised, controlled investigator blinded, crossover design is being used. Participants will be reviewed at 3 and 6 months. Couples will be randomised to start either with latex condoms alone (Durex Extra Safe) or with additional Duragel (nonoxynol-9 contracceptive gel) applied to the outside of the condom prior to initial penetration. Participants are heterosexual couples using condoms for vaginal non-commercial intercourse in stable relationships of at least 3 months duration. Those under 18, or unable to provide data due to communication difficulties will be excluded from the trial.

Data will be collected by questionnaires for all subjects on their contraceptive and STI history, key demographic, social and behavioural factors relevant to condom failure risk at baseline. At crossover and trial end the rate and types of condom failure, side effects and acceptability of additional spermicide, and health service and subject costs are collected. A random sample of subjects also participate in a detailed semi-structured interview at the end of the study, covering their recent experiences of condom failure, and opinions about condoms in general, including the use of additional spermicide. These qualitative findings will then be discussed in patient and professional focus groups as a proxy for respondent checking and data triangulation.

The research will provide valuable, detailed information on factors associated with condom failure. Confirmation of the previous finding of the protective effects of additional spermicide would have a potentially major international impact in the fields of family planning and infectious diseases.

ELIGIBILITY:
Inclusion Criteria:

* Condom using heterosexual couples in stable relationships

Exclusion Criteria:

* Allergy to latex and or nonoxynol-9, communication difficulties precluding data collection

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200
Dates: Start 1998-04; Study Completion 2002-04

PRIMARY OUTCOMES:
Condom failure- breakage or slippage

CONTACTS AND LOCATIONS:
Overall Officials: Mark B Gabbay, MBChG MD, Principal Investigator — University of Liverpool

REFERENCES:
- [Background] Gabbay M, Thomas J. When free condoms and spermicide are not enough: barriers and solutions to participant recruitment to community-based trials. Control Clin Trials. 2004 Aug;25(4):388-99. doi: 10.1016/j.cct.2004.06.004. PMID 15296813
- [Derived] Gabbay MB, Thomas J, Gibbs A, Hold P. A randomized crossover trial of the impact of additional spermicide on condom failure rates. Sex Transm Dis. 2008 Oct;35(10):862-8. doi: 10.1097/OLQ.0b013e31817fb802. PMID 18685543